CLINICAL TRIAL: NCT05527067
Title: A Registered Observational Cohort Study on α-Synucleinopathy
Brief Title: A Registered Cohort Study on α-Synucleinopathy
Status: Recruiting | Type: Observational
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Cohort-PDS
Record Dates: First submitted 2022-08-28; First posted 2022-09-02 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2022-08

CONDITIONS: α-synucleinopathy
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- α-synucleinopathy: Participants with clinical diagnosis of α-synucleinopathy.
  Interventions: Other: Data collection
- Healthy controls: Healthy controls
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Neuropsychological assessment, brain MRI, electroencephalogram and biomarker datas will be collected
  Groups: α-synucleinopathy
Other: Data collection — Neuropsychological assessment, brain MRI, electroencephalogram and biomarker datas will be collected
  Groups: Healthy controls

SUMMARY:
α-Synucleinopathy is a cluster of neurodegenerative disease with motor and non-motor symptom. The data to be collected is intended to help healthcare providers make important medical decisions concerning α-synucleinopathy, through an enhanced understanding of the natural history, progression and multi-omics datasets of α-synucleinopathy.

DETAILED DESCRIPTION:
α-Synucleinopathy is a cluster of neurodegenerative disease with motor and non-motor symptom, including Parkinson's disease (PD), multiple system atrophy (MSA) and dementia with lewy bodies (DLB). The data to be collected is intended to help healthcare providers make important medical decisions concerning α-synucleinopathy, through an enhanced understanding of the natural history, progression and multi-omics datasets of α-synucleinopathy. Datas will be accumulated retrospectively at research entry and prospectively during follow up.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a clinical diagnosis of primary α-synucleinopathy
* Unrelated healthy controls

Exclusion Criteria:

* Patients with secondary α-synucleinopathy that cannot be excluded.
* Patients with other neurological disorders.
* Pregnant or lactating women.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with a clinical diagnosis of PD, DLB and MSA.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
UPDRS /UMSARS scores | Baseline
  Disease severity was evaluated by the neurologist using the united Parkinson's disease rating scale (UPDRS) or united multiple system atrophy rating scale (UMSARS) separately as diagnosed.

SECONDARY OUTCOMES:
H&Y stage | Baseline
  The Hoehn and Yahr （H&Y)
MoCA scores | Baseline
  The Montreal Cognitive Assessment (MoCA)
ACE-III scores | Baseline
  Addenbrooke's Cognitive Examination (ACE) score
Mean arterial pressure after 3 minutes of upright posture versus decubitus position (mmHg) | Baseline
  Mean arterial pressure was calculated as ⅓ pulse pressure + diastolic pressure.
HRV (ms) | Baseline
  Heart rate variability (HRV) was calculated as the maximum bpm - minimum bpm.
Plasma α-synuclein levels (ng/ml) | Baseline
Vic | Baseline
  The intra-cellular compartment (Vic) of the Neurite Orientation Dispersion and Density Imaging (NODDI) model represents diffusion within the axons and cells.
PAF (Hz) | Baseline
  The alpha-peak frequency (PAF) is the frequency with the highest power within the alpha-band.
Vic | 1 year after Baseline
  The intra-cellular compartment (Vic) of the Neurite Orientation Dispersion and Density Imaging (NODDI) model represents diffusion within the axons and cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No